CLINICAL TRIAL: NCT00000911
Title: An Observational Study of Subjects With Primary HIV Infection: A Study of the UCSD Acute/Early HIV Infection (AEHIV) Clinical Studies Unit
Brief Title: A Study to Monitor Patients With Primary or Early HIV Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Rona Siskind, DAIDS
Other Study IDs: AI-05-001; SD AEHIV 001; AEHIV 001; AIEDRP AI-05-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: HIV Infections
Keywords: Semen; HIV-1; Immunity, Cellular; Lymph Nodes; Viremia; Antibodies, Viral; Vagina; Viral Load; Acute Infection
MeSH Terms: conditions — HIV Infections; Viremia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, lymph node tissue, CSF, and semen or vaginal secretion specimens

SUMMARY:
The purpose of this study is to monitor patients who recently have been infected with HIV in order to learn how their immune systems respond to HIV infection and to study how the virus acts in their bodies.

Primary HIV infection occurs within 20 days to 8 weeks following exposure to HIV. The symptoms of primary HIV infection are usually fever, tiredness, headache, or muscle aches. However, symptoms vary greatly from person to person, and some people might not experience any symptoms at all. Because these symptoms also resemble the cold or the flu, it is difficult to identify patients with primary HIV infection. Information gathered from this study will help doctors decide what kind of treatment is best to give patients who recently have been infected.

DETAILED DESCRIPTION:
Primary HIV-1 infection is frequently identified as a nonspecific viral syndrome occurring within 20 days to 8 weeks following a documented HIV exposure. However, symptoms vary from person to person, and some people undergo asymptomatic seroconversion. Because of the difficulty identifying patients with either acute HIV infection (within 30 days of initial infection) or early infection (within 12 months of initial infection), no systematic review of viral dynamics or immunodynamics in this patient population has been undertaken. A better understanding of the virologic and immunologic parameters during acute and early HIV infection should provide information relevant to the optimal design of future clinical therapeutic trials.

The only patient intervention is obtaining blood, lymph node tissue, CSF, and semen or vaginal secretion specimens at designated intervals according to the schedule of evaluations. Patients are followed for 5 years. Patients may elect to start or discontinue antiretroviral therapy at any time; however, no antiretroviral therapy is administered as part of this study. Descriptive analysis includes tolerance and toxicity, magnitude and durability of RNA suppression, magnitude and durability of immunologic responses (CD4 and CD8 cells), and decay and emergence of resistant virus in tissue reservoirs (CSF, genital secretions, and lymph nodes).

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old (consent of parent or guardian required if under 18).
* Have acute or early HIV infection. The stage of HIV infection will depend on the results of certain lab tests.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have recently been infected with HIV
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 1999-10; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Little, Principal Investigator; Diane Havlir, Principal Investigator
Locations (1):
- University of California, San Diego, San Diego, California, United States